# Calistar A vs. Calistar S - Comparative Cohort Retrospective Analysis of Single Incision POP Systems

ID: CaSCaA

Version number: Ver\_03
Date: 28/05/2018

NCT03715803

**Study Protocol** 

Version 03 28/05/2018 Pag. **1** of **7** 

#### CALISTAR A VS CALISTAR S – COHORT RETROSPECTIVE ANALYSIS

(Ver\_03 - 28/05/2018)

#### PROTOCOL APPROVAL

| Responsible/Protocol Author/PI | (dd/mm/yyyy) |
|--------------------------------|--------------|

This protocol has been designed in accordance with the principles of Good Clinical Practices, EN-ISO 14155, Declaration of Helsinki and other applicable regulatory requirements.

Version 03 28/05/2018 Pag. **2** of **7** 

#### SIGNATURE PAGE

#### CALISTAR A VS CALISTAR S – COHORT RETROSPECTIVE ANALYSIS

(Ver\_03 - 28/05/2018)

I have read this protocol and agree to adhere to the requirements. I will provide copies of this protocol and all pertinent information to the study personnel under my supervision and my hospital ethics committee / institutional review board (EC/ORB). I will discuss this material with them and ensure they are fully informed regarding the device and the conduct of the study according to this protocol, applicable laws, and applicable regulatory requirements including Good Clinical Practices.

| | Clinical Site Name | |
|---------------------------------------|--------------------|------|
| Cita Daireira Havastiastas Ciastus | | |
| Site Principal Investigator Signature | | Date |

Version 03 28/05/2018 Pag. **3** of **7** 

## TABLE OF CONTENTS

| SIGNATURE PAGE | 3 |
|---------------------|---|
| Table of contents | 4 |
| GENERAL INFORMATION | 5 |
| RIRI IOGRAPHY | 7 |

### **GENERAL INFORMATION**

| Protocol ID | |
|---|---|
| Short title | CALISTAR A VS CALISTAR S – Cohort retrospective analysis |
| EudraCT number | N/a |
| Version | 3.0 |
| Date | 28/05/2018 |
| Coordinating investigator/project leader | Dr. A. Sampietro, Gynecologist |
| | Hospital Universitario Austral, Department of gynaecology |
| | Av. Juan Domingo Perón 1500, Pilar Centro, Buenos Aires, |
| | Argentina |
| | + 54-230-448-2163 |
| | asampietro@live.com.ar |
| Principal investigators | See Annex 1 |
| Sponsor | N/a |
| Product | Calistar A and Calistar S Single Incision POP System from |
| | Promedon. The products which are the object of this study have |
| | the approval according the CE-Guideline 93/42/EWG. |
| Objective | To compare the initial outcomes and complication of a high |
| | weight and a low weight meshes, Calistar A and Calistar S, |
| | respectively, implanted through a single incision to treat anterior |
| | and apical prolapses. |
| Study design | Multicentre, post-market, retrospective, two arms, non- |
| | randomized comparative study. |
| Study population | Adult female |
| Main study parameters/ primary | Effectiveness of Calistar S and Calistar A will be assessed by cure |
| endpoints | criteria of Barber, that is: |
| | - Lowest point of POP-Q < 0 (no points beyond the hymen) |
| | - No subjective bothersome symptoms (absence of vaginal bulge |
| | symptoms) |
| | - No re-treatment/interventions on year post procedure. |

Version 03 28/05/2018 Pag. **5** of **7** 

| Secondary endpoints | The secondary endpoint is defined as the objective assessment of |
|---|---|
| | POP by POP-Q. POP-Q staging will be compared pre- and post- |
| | operative. |
| | The subjective outcome is defined as the assessment of |
| | subjective symptoms resulting from POP by validated quality of |
| | life (QoL) questionnaires (improvement of the QoL of the subjects |
| | compared to the baseline values): |
| | - Pelvic Floor Distress Inventory (PFDI 20) to assess the impact of |
| | urinary, prolapse and colorectal distress post-operative. |
| | - Pelvic Organ Prolapse/ Urinary Incontinence Sexual |
| | Questionnaire (PISQ-12) to evaluate sexual function in women |
| | with pelvic organ prolapse and/or urinary incontinence post- |
| | operative. |
| | - Patient Global Impression to evaluate patient satisfaction with |
| | the experience and the result of procedure. |
| | Type of surgery and operative time will be compared for both |
| | pelvic floor systems repair. |
| Safety endpoints | Operative complications such as bladder injury and blood loss will |
| | be evaluated. Complications related to the use of meshes such as |
| | vaginal pain, infection and mesh erosion will be assessed. |
| Inclusion criteria | Female; |
| | Anterior and apical prolapse Stage 3 (according to POP-Q) or |
| | more with or without SUI; |
| | Primary or recurrent treatment with Calistar S or Calistar A; |
| | At least 6 months follow-up |
| Exclusion criteria | Recurrent vaginal infections; |
| | Chronic colorectal diseases (chronic nonspecific ulcerative colitis, |
| | diverticulitis, diverticulosis, Chron's disease, irritable bowel |
| | syndrome, familial polyposis); |
| | Presence of any coagulopathies; |
| | Impairment of the immune system or any condition that |
| | compromises recovery; |
| | Prior irradiation; |
| | Chronic pelvic pain |

Version 03 28/05/2018 Pag. **6** of **7** 

#### **BIBLIOGRAPHY**

- 1. SCENIHR. Opinion on The safety of surgical meshes used in urogynecological surgery. 2015. 105 p.
- 2. Amid PK. Classification of biomaterials and their related complications in abdominal wall hernia surgery. Hernia [Internet]. 1997;1(1):15–21. Available from: http://link.springer.com/10.1007/BF02426382
- 3. De Tayrac R, Madelenat P. Évolution Des DiffRentes Voies D'Abord Chirurgicales Dans L'Incontinence Urinaire D'Effort ÉMinine. Gynecol Obstet Fertil. 2004;32(12):1031–8.
- 4. PALMA P, RICCETTO C, ALTUNA S, BARREIRO TM, SARDI J, LEDESMA M, et al. Simultaneous single incision transvaginal mesh to treat anterior and apical prolapses A midterm results. IUGA 38th Annu Meet. 2013;Poster 470.
- 5. Bigozzi MA, Provenzano S, Maeda F, Palma PCR, Riccetto CZ. In Vivo Biomechanical Properties of Heavy Versus Light Weight Monofilament Polypropylene Meshes. Does the Knitting Pattern Matter? Neurourol Urodyn. 2015;
- 6. Barber MD, Brubaker L, Nygaard I, Wheeler TL, Schaffer J, Chen Z, et al. Defining success after surgery for pelvic organ prolapse. Obstet Gynecol. 2009;114(3):600–9.
- 7. Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, et al. an International Urogynecological Association (luga) / International Continence Society (lcs) Joint Report on the Terminology for Female Pelvic Organ Prolapse (Pop) . 2015;655–84.
- 8. Toozs-Hobson P, Freeman RM, Barber M, Maher C, Haylen B, Athanasiou S, et al. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for reporting outcomes of surgical procedures for pelvic organ prolapse. Int Urogynecol J. 2012;23(5):527–35.
- 9. Clavien P a, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, et al. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009;250(2):187–96.

Version 03 28/05/2018 Pag. **7** of **7**